CLINICAL TRIAL: NCT05972785
Title: Association of Long-term Use of Calcium Channel Blockers (CCB) and Risk of Breast Cancer: A Retrospective Longitudinal Observational Study
Brief Title: Long-term Use of CCB and Breast Cancer Risk
Status: Active, not recruiting | Type: Observational
Sponsor: Curtin University (Other)
Responsible Party: Principal Investigator, Rachael Moorin, Professor, Curtin University
Other Study IDs: 2014896
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hypertension,Essential; Breast Cancer
MeSH Terms: conditions — Essential Hypertension; Breast Neoplasms | interventions — Calcium Channel Blockers; Adrenergic beta-Antagonists; Diuretics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- No AHT: Women with HTN with no AHT use
  Interventions: Drug: None AHT
- AHT but non-CCB: Women with HTN exposed to other antihypertensive medicines but not exposed to calcium channel blockers
  Interventions: Drug: Beta blocker; Drug: Diuretic; Drug: RAS; Drug: Other AHT
- CCB only: Women with HTN exposed to calcium channel blockers but not exposed to other antihypertensive medicines
  Interventions: Drug: Calcium channel blocker
- Both CCB and non-CCB: Women with HTN exposed to both calcium channel blockers and other antihypertensive medicines.
  Interventions: Drug: Calcium channel blocker; Drug: Beta blocker; Drug: Diuretic; Drug: RAS; Drug: Other AHT

INTERVENTIONS:
Drug: Calcium channel blocker — Drugs with ATC code C08 will be categorised as calcium channel blockers.
  Groups: Both CCB and non-CCB; CCB only
Drug: Beta blocker — Drugs with ATC code C07 will be categorised as beta-blockers.
  Groups: AHT but non-CCB; Both CCB and non-CCB
Drug: Diuretic — Drugs with ATC code C03 will be categorised as diuretics.
  Groups: AHT but non-CCB; Both CCB and non-CCB
Drug: RAS — Drugs with ATC code C09 will be categorised as RAS (agents acting on the renin angiotensin system).
  Groups: AHT but non-CCB; Both CCB and non-CCB
Drug: Other AHT — Drugs with ATC code C02 will be categorised as other antihypertensives.
  Groups: AHT but non-CCB; Both CCB and non-CCB
Drug: None AHT — None AHT
  Groups: No AHT

SUMMARY:
The goal of this retrospective observational study is to examine whether long-term calcium channel blocker (CCB) use is associated with the development of breast cancer amongst women enrolled in three longitudinal cohort studies in Australia and the Netherlands . The main questions it aims to answer are:

* Is long-term CCB use associated with the development of breast cancer amongst women enrolled in three longitudinal cohort studies in Australia and the Netherlands and what is the dose-response nature of this association.
* Does differences in the association between calcium channel blocker use and the development of breast cancer exist between Australian and Dutch women.

The investigators will utilise data from the Australian Longitudinal Study on Women's Health (ALSWH) , 45 and Up Study and Rotterdam study.

DETAILED DESCRIPTION:
Aims: To examine the association between long-term calcium channel blocker (CCB) use and the development of breast cancer.

Data sources: the Australian Longitudinal Study on Women's Health , 45 and Up Study, Rotterdam study and linked administrative data.

Study cohort: Women with self-reported hypertension (HTN) without prior breast cancer.

Harmonisation: Relevant variables will be checked for harmonisation in which variables available in all three cohort will be used in the harmonised analysis. The variables will be checked on the definition, measurement and harmonisation rules. Variables that cannot be harmonised across the cohorts will be used in the cohort specific analyses.

Exposure measurement: The primary exposure is the use of CCB, which will be identified by the anatomical therapeutic chemical code (C08) in the medicine data. Exposure to CCB as well as other antihypertensive (AHT) medicines will be captured separately as the cumulative dose-duration of exposure during follow up. Participants will be stratified in four groups: women with HTN with no AHT use, women with HTN exposed to CCB only, women with HTN exposed to non-CCB and women with HTN exposed to both CCB and non-CCB.

Outcome measurement: Data on a diagnosis of invasive breast cancer will be obtained from cancer registries and hospital admission data using ICD-10 code of C50.x.

Potential confounders: age, education, marital status, socioeconomic status, body mass index, diabetes, heart disease, stroke, age when had first child, parity, history of hysterectomy or oophorectomy, use of hormonal contraception, use of hormonal replacement therapy.

Statistical analysis: The association between CCB use and breast cancer risk will be estimated by the Fine and Gray competing risk regression model in which a first diagnosis of invasive breast cancer will be treated as the principle event and death and bilateral mastectomy (without a diagnosis of breast cancer) will be competing risks. The nonlinear threshold models will be used to capture any differential effect of the cumulative dose-duration of CCB while simultaneously accounting for the cumulative dose-duration of other AHT exposure on breast cancer risk. Other confounders will be accounted for in the models using propensity scores.

Implications: Results from this study will contribute to addressing the concerns about using CCB for hypertension treatment in women, particularly in those who have high risk of breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Alive and still enrolled in the longitudinal cohort at the study entry (2004 to 2009)
* Self-reported/diagnosed hypertension at study entry.

Exclusion criteria:

+ A history of breast cancer.

Min Age: 45 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will include eligible women enrolled in three longitudinal cohorts: ALSWH, 45 and Up Study and the Rotterdam study.
Sampling Method: Probability Sample
Enrollment: 68500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incident rate of invasive breast cancer | From cohort entry until the earliest date of one of the following: a diagnosis of invasive breast cancer, bilateral mastectomy (without breast cancer) or death, assessed up to 14 years.
  The outcome will be defined based on the ICD-10 code of C50.x (malignant neoplasm of breast).

CONTACTS AND LOCATIONS:
Locations (1):
- Curtin university, Bentley, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho C, Ha NT, Youens D, Abhayaratna WP, Bulsara MK, Hughes JD, Mishra G, Pearson SA, Preen DB, Reid CM, Ruiter R, Saunders CM, Stricker BH, van Rooij FJA, Wright C, Moorin R. Association between long-term use of calcium channel blockers (CCB) and the risk of breast cancer: a retrospective longitudinal observational study protocol. BMJ Open. 2024 Mar 8;14(3):e080982. doi: 10.1136/bmjopen-2023-080982. PMID 38458796